CLINICAL TRIAL: NCT05425394
Title: A Study of Effects of Delay in the First Bathing Time of Newborns on the Rate of Body Temperature and the Rate of Exclusive Breastfeeding: A Randomized Controlled Trial
Brief Title: A Study of Effects of Delay in the First Bathing Time of Body Temperature and the Rate of Exclusive Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Di-Ling Huang, Head nursing, Cardinal Tien Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DHuang-0001
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Newborn Hypothermia
Keywords: delayed bathing; body temperature; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed first bath time (Experimental): Delay first bath to 8 hours after birth
  Interventions: Behavioral: Delay first bath
- regular bath (No Intervention): Birth temperature 36.5°C, regular bath

INTERVENTIONS:
Behavioral: Delay first bath — Newborns delay first bath to 8 hours after birth
  Arms: delayed first bath time

SUMMARY:
Using delaying the first bathing by 8 hours as an interventional measure, considering the consistent effect of physiological maturity, newborns with a gestational age of ≥37 weeks were selected as the subjects in the nursery cases, and randomly assigned to the delayed bathing group and the routine bathing group , 10 minutes before bathing, immediately after bathing, 10 minutes, 30 minutes, and 60 minutes to analyze the differences in body temperature of the cases, and the differences in the rate of exclusive breastfeeding at discharge.

DETAILED DESCRIPTION:
The subjects of this study came from newborn babies in the nursery of a teaching hospital in the northern region. The research design was reviewed and approved by the Human Trials Committee. Can freely choose whether to participate in the research project or withdraw, willing participants to inform the research project and fill in the consent form and basic information form, inform that they can withdraw at any time during the research period, and divide the participating infants into the experimental group and the control group through a random allocation form , after the newborn arrives in the baby room, the nursing staff will evaluate the newborn, and then perform an oil bath with baby oil to remove the fetal fat on the body, and then follow the newborn bathing procedure of our hospital. Wash the whole body with water, about 1-2 hours after birth; the control group took the first bath as usual; the experimental group postponed the last step of washing the whole body after washing the face and head to 8 hours after birth , personnel must wear gloves to take care of newborns before bathing. The bathing process was performed by nurses in the baby room. Body temperature was measured 10 minutes before, immediately after, 10 minutes, 30 minutes, and 60 minutes after bathing, and the exclusive breastfeeding situation at the time of discharge was counted. After all measurements are completed, a 100 yuan supermarket coupon will be given.

ELIGIBILITY:
Inclusion Criteria:

* Apparently normal newborn with status ranging from normal to good
* mean gestational age ≥37 weeks
* birth weight ≥2500 g
* Apgar score of at least 7 within 1-5 minutes
* birth rectal temperature ≥36.5°C
* without any major change or signs or symptoms of sepsis.

Exclusion Criteria:

* The mother is younger than 20 years old
* has recently had symptoms of fever, leukocytosis, respiratory tract infection or urinary tract infection
* the mother has diseases such as diabetes, hyperthyroidism, and a positive history of type B streptococcus or other blood and body fluid infectious diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
body temperature after bath | temperature measurement : 10 minutes after bathing
  The degree of decrease in body temperature after bathing compared to before bathing

SECONDARY OUTCOMES:
Exclusive breastfeeding rate | 3 to 5 days
  Neonatal feeding methods during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- DiLing Huang, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study is a personal research project, and the subject's instructions and consent form for human trials inform the subjects that the data in the study is for this study only.

REFERENCES:
- [Background] Wang Yating, Wang Xiuhe, Wu Sujin, Zheng Yufang, Liao Wenling (2014). A study on the choice of feeding method and its related factors in parturients. Joseph Medical Journal, 8(1), 5-16.
- [Background] Lin Yujing, Yang Jialing, Gao Meihua, Li Jingyi (2012). Correlation between perinatal breastfeeding instruction and maternal practice of 24-hour parent-child rooming. Chang Gung Nursing, 23(1), 27-40.
- [Background] Lin YW, Tzeng YL, Yang YL. [Mother-friendly childbirth practices and breastfeeding]. Hu Li Za Zhi. 2013 Feb;60(1):5-10. doi: 10.6224/JN.60.1.5. Chinese. PMID 23386519
- [Background] Ke Huijuan, Zhong Yulun, Chen Shufen (2019). A retrospective cohort study on the effect of continuous exclusive breastfeeding on the 24-hour parent-child rooming strategy in a medical center. Rong Total Nursing, 36(4), 343-352.
- [Background] Xu Yufen, Liu Xinyi, Li Zhaohui, Chen Shujuan (2010). Improvement programs to reduce the incidence of neonatal hypothermia. Journal of Midwifery, 52, 93-104.
- [Background] Gao Yuxiu, Li Fengxue, and Wang Guoming (2012). Influence of primipara background factors on breastfeeding experience and self-efficacy. Journal of Midwifery, 54, 56-67.
- [Background] Chen Guanying, Wei Ziyi, Huang Xiaoyu, Xu Yunxin (2019). A project to improve hypothermia for neonates admitted to the moderate-severe ward in the delivery room. Journal of Nursing, 66(4), 71-78.
- [Background] You Shuzhen (2018). Discussion on the related factors of continuous breastfeeding in postpartum women.
- [Background] Ye Jinxue (2015). The Guardianship of Successful Breastfeeding. Taiwan Medicine, 19(6), 643-649.
- [Background] Anderson J. An Organization-Wide Initiative to Implement Parent-Performed, Delayed Immersion Bathing. Nurs Womens Health. 2021 Feb;25(1):63-70. doi: 10.1016/j.nwh.2020.11.006. Epub 2021 Jan 13. PMID 33450241
- [Background] Association of Women's Health, Obstetric and Neonatal Nurses. （2018）. Neonatal skin care: Evidence-based clinical practice guideline （4th ed.）. AWHONN.
- [Background] Bhutta ZA, Das JK, Bahl R, Lawn JE, Salam RA, Paul VK, Sankar MJ, Blencowe H, Rizvi A, Chou VB, Walker N; Lancet Newborn Interventions Review Group; Lancet Every Newborn Study Group. Can available interventions end preventable deaths in mothers, newborn babies, and stillbirths, and at what cost? Lancet. 2014 Jul 26;384(9940):347-70. doi: 10.1016/S0140-6736(14)60792-3. Epub 2014 May 19. PMID 24853604
- [Background] Binns C, Lee MK, Kagawa M. Ethical Challenges in Infant Feeding Research. Nutrients. 2017 Jan 11;9(1):59. doi: 10.3390/nu9010059. PMID 28085057
- [Background] Bissinger RL, Annibale DJ. Thermoregulation in very low-birth-weight infants during the golden hour: results and implications. Adv Neonatal Care. 2010 Oct;10(5):230-8. doi: 10.1097/ANC.0b013e3181f0ae63. PMID 20838071
- [Background] Blackburn, S. T., （2003）. Thermoregulation. In S. T. Blackburn （Ed.）, Maternal, fetal, & neonatal physiology: A clinical perspective （2nd ed., pp. 707-730）. Philadelphia, Saunders.
- [Background] Bowden, V. R., & Greenberg, C. S. （2010）. Children and their families: The continuum of care. Lippincott Williams & Wilkins.
- [Background] Lund CH, Osborne JW, Kuller J, Lane AT, Lott JW, Raines DA. Neonatal skin care: clinical outcomes of the AWHONN/NANN evidence-based clinical practice guideline. Association of Women's Health, Obstetric and Neonatal Nurses and the National Association of Neonatal Nurses. J Obstet Gynecol Neonatal Nurs. 2001 Jan-Feb;30(1):41-51. PMID 11277161
- [Background] Brogan J, Rapkin G. Implementing Evidence-Based Neonatal Skin Care With Parent-Performed, Delayed Immersion Baths. Nurs Womens Health. 2017 Dec;21(6):442-450. doi: 10.1016/j.nwh.2017.10.009. PMID 29223208
- [Background] Byaruhanga R, Bergstrom A, Okong P. Neonatal hypothermia in Uganda: prevalence and risk factors. J Trop Pediatr. 2005 Aug;51(4):212-5. doi: 10.1093/tropej/fmh098. Epub 2005 May 25. PMID 15917265
- [Background] Medoff Cooper B, Holditch-Davis D, Verklan MT, Fraser-Askin D, Lamp J, Santa-Donato A, Onokpise B, Soeken KL, Bingham D. Newborn clinical outcomes of the AWHONN late preterm infant research-based practice project. J Obstet Gynecol Neonatal Nurs. 2012 Nov-Dec;41(6):774-85. doi: 10.1111/j.1552-6909.2012.01401.x. Epub 2012 Aug 3. PMID 22861492
- [Background] Crenshaw JT. Healthy Birth Practice #6: Keep Mother and Baby Together- It's Best for Mother, Baby, and Breastfeeding. J Perinat Educ. 2014 Fall;23(4):211-7. doi: 10.1891/1058-1243.23.4.211. PMID 25411542
- [Background] DiCioccio HC, Ady C, Bena JF, Albert NM. Initiative to Improve Exclusive Breastfeeding by Delaying the Newborn Bath. J Obstet Gynecol Neonatal Nurs. 2019 Mar;48(2):189-196. doi: 10.1016/j.jogn.2018.12.008. Epub 2019 Jan 21. PMID 30677407
- [Background] DiGirolamo AM, Grummer-Strawn LM, Fein SB. Effect of maternity-care practices on breastfeeding. Pediatrics. 2008 Oct;122 Suppl 2:S43-9. doi: 10.1542/peds.2008-1315e. PMID 18829830
- [Background] Eidelman AI. Breastfeeding and the use of human milk: an analysis of the American Academy of Pediatrics 2012 Breastfeeding Policy Statement. Breastfeed Med. 2012 Oct;7(5):323-4. doi: 10.1089/bfm.2012.0067. Epub 2012 Sep 4. No abstract available. PMID 22946888
- [Background] Fernandez D, Antolin-Rodriguez R. Bathing a Premature Infant in the Intensive Care Unit: A Systematic Review. J Pediatr Nurs. 2018 Sep-Oct;42:e52-e57. doi: 10.1016/j.pedn.2018.05.002. Epub 2018 May 18. PMID 29779763
- [Background] Gardner, S. L., Carter, B. S., Enzman-Hines, M. I., & Niermeyer, S. （2020）. Merenstein & Gardner's Handbook of Neonatal Intensive Care-E-Book: An Interprofessional Approach. Elsevier Health Sciences.
- [Background] George S, Phillips K, Mallory S, Holmquistova I, Hare R, Allen S, Higgins M, Shapiro SE. A pragmatic descriptive study of rewarming the newborn after the first bath. J Obstet Gynecol Neonatal Nurs. 2015 Mar-Apr;44(2):203-9. doi: 10.1111/1552-6909.12556. Epub 2015 Feb 24. PMID 25712473
- [Background] Hackman PS. Recognizing and understanding the cold-stressed term infant. Neonatal Netw. 2001 Dec;20(8):35-41. doi: 10.1891/0730-0832.20.8.35. PMID 12144102
- [Background] Hughes Driscoll CA, Pereira N, Lichenstein R. In-hospital Neonatal Falls: An Unintended Consequence of Efforts to Improve Breastfeeding. Pediatrics. 2019 Jan;143(1):e20182488. doi: 10.1542/peds.2018-2488. PMID 30593451
- [Background] Kelly PA, Classen KA, Crandall CG, Crenshaw JT, Schaefer SA, Wade DA, Cramer MN, Aryal S, Fossee KR. Effect of Timing of the First Bath on a Healthy Newborn's Temperature. J Obstet Gynecol Neonatal Nurs. 2018 Sep;47(5):608-619. doi: 10.1016/j.jogn.2018.07.004. Epub 2018 Aug 8. PMID 30096281
- [Background] Knobel, R. B., （2014）. Fetal and neonatal thermal physiology. Newborn and Infant Nursing Reviews, 14（2）, 45-49.
- [Background] Koopman I, Callaghan-Koru JA, Alaofin O, Argani CH, Farzin A. Early skin-to-skin contact for healthy full-term infants after vaginal and caesarean delivery: a qualitative study on clinician perspectives. J Clin Nurs. 2016 May;25(9-10):1367-76. doi: 10.1111/jocn.13227. Epub 2016 Mar 30. PMID 27027262
- [Background] Kuller, J. M., （2014）. Update on newborn bathing. Newborn and Infant Nursing Reviews, 14（4）, 166-170.
- [Background] Laptook AR, Salhab W, Bhaskar B; Neonatal Research Network. Admission temperature of low birth weight infants: predictors and associated morbidities. Pediatrics. 2007 Mar;119(3):e643-9. doi: 10.1542/peds.2006-0943. Epub 2007 Feb 12. PMID 17296783
- [Background] Laptook A, Jackson GL. Cold stress and hypoglycemia in the late preterm ("near-term") infant: impact on nursery of admission. Semin Perinatol. 2006 Feb;30(1):24-7. doi: 10.1053/j.semperi.2006.01.014. PMID 16549210
- [Background] Liberth, M., & Fontana, J. （2018）. Benefits of Delayed Bathing. Journal of Obstetric, Gynecologic & Neonatal Nursing, 47（3）, S30-S31
- [Background] Lipka, D. V., & Schulz, M. K. （2012）. "Wait for eight": Improvement of newborn outcomes by the implementation of newborn bath delay. Journal of Obstetric, Gynecologic, & Neonatal Nursing, 41（s1）, S46-S47.
- [Background] Lund C. Bathing and Beyond: Current Bathing Controversies for Newborn Infants. Adv Neonatal Care. 2016 Oct;16 Suppl 5S:S13-S20. doi: 10.1097/ANC.0000000000000336. PMID 27676109
- [Background] Lunze K, Bloom DE, Jamison DT, Hamer DH. The global burden of neonatal hypothermia: systematic review of a major challenge for newborn survival. BMC Med. 2013 Jan 31;11:24. doi: 10.1186/1741-7015-11-24. PMID 23369256
- [Background] Mardini J, Rahme C, Matar O, Abou Khalil S, Hallit S, Fadous Khalife MC. Newborn's first bath: any preferred timing? A pilot study from Lebanon. BMC Res Notes. 2020 Sep 14;13(1):430. doi: 10.1186/s13104-020-05282-0. PMID 32928289
- [Background] Merazzi D, Bresesti I, Tagliabue P, Valsecchi MG, De Lorenzo P, Lista G; Collaboration Group. Body temperature at nursery admission in a cohort of healthy newborn infants: results from an observational cross-sectional study. Ital J Pediatr. 2020 Apr 15;46(1):46. doi: 10.1186/s13052-020-0810-z. PMID 32293526
- [Background] Merten S, Dratva J, Ackermann-Liebrich U. Do baby-friendly hospitals influence breastfeeding duration on a national level? Pediatrics. 2005 Nov;116(5):e702-8. doi: 10.1542/peds.2005-0537. PMID 16263985
- [Background] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Background] Hellwig JP. Providing evidence-based care: ANA launches research toolkit. Nurs Womens Health. 2011 Dec;15(6):545-6. doi: 10.1111/j.1751-486X.2011.01688.x. No abstract available. PMID 22900697
- [Background] Ng CA, Ho JJ, Lee ZH. The effect of rooming-in on duration of breastfeeding: A systematic review of randomised and non-randomised prospective controlled studies. PLoS One. 2019 Apr 25;14(4):e0215869. doi: 10.1371/journal.pone.0215869. eCollection 2019. PMID 31022227
- [Background] Patel A, Bucher S, Pusdekar Y, Esamai F, Krebs NF, Goudar SS, Chomba E, Garces A, Pasha O, Saleem S, Kodkany BS, Liechty EA, Kodkany B, Derman RJ, Carlo WA, Hambidge K, Goldenberg RL, Althabe F, Berrueta M, Moore JL, McClure EM, Koso-Thomas M, Hibberd PL. Rates and determinants of early initiation of breastfeeding and exclusive breast feeding at 42 days postnatal in six low and middle-income countries: A prospective cohort study. Reprod Health. 2015;12 Suppl 2(Suppl 2):S10. doi: 10.1186/1742-4755-12-S2-S10. Epub 2015 Jun 8. PMID 26063291
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal Resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S204-41. doi: 10.1161/CIR.0000000000000276. No abstract available. PMID 26472855
- [Background] Perlman J, Kjaer K. Neonatal and Maternal Temperature Regulation During and After Delivery. Anesth Analg. 2016 Jul;123(1):168-72. doi: 10.1213/ANE.0000000000001256. PMID 27314693
- [Background] Preer G, Pisegna JM, Cook JT, Henri AM, Philipp BL. Delaying the bath and in-hospital breastfeeding rates. Breastfeed Med. 2013 Dec;8(6):485-90. doi: 10.1089/bfm.2012.0158. Epub 2013 May 2. PMID 23635002
- [Background] Rito AI, Buoncristiano M, Spinelli A, Salanave B, Kunesova M, Hejgaard T, Garcia Solano M, Fijalkowska A, Sturua L, Hyska J, Kelleher C, Duleva V, Music Milanovic S, Farrugia Sant'Angelo V, Abdrakhmanova S, Kujundzic E, Peterkova V, Gualtieri A, Pudule I, Petrauskiene A, Tanrygulyyeva M, Sherali R, Huidumac-Petrescu C, Williams J, Ahrens W, Breda J. Association between Characteristics at Birth, Breastfeeding and Obesity in 22 Countries: The WHO European Childhood Obesity Surveillance Initiative - COSI 2015/2017. Obes Facts. 2019;12(2):226-243. doi: 10.1159/000500425. Epub 2019 Apr 26. PMID 31030194
- [Background] Ruschel LM, Pedrini DB, Cunha MLCD. Hypothermia and the newborn's bath in the first hours of life. Rev Gaucha Enferm. 2018 Oct 22;39:e20170263. doi: 10.1590/1983-1447.2018.20170263. English, Portuguese. PMID 30365754
- [Background] Russo A, McCready M, Torres L, Theuriere C, Venturini S, Spaight M, Hemway RJ, Handrinos S, Perlmutter D, Huynh T, Grunebaum A, Perlman J. Reducing hypothermia in preterm infants following delivery. Pediatrics. 2014 Apr;133(4):e1055-62. doi: 10.1542/peds.2013-2544. Epub 2014 Mar 31. PMID 24685958
- [Background] SILVERMAN WA, FERTIG JW, BERGER AP. The influence of the thermal environment upon the survival of newly born premature infants. Pediatrics. 1958 Nov;22(5):876-86. No abstract available. PMID 13600915
- [Background] Singh G, Archana G. Unraveling the mystery of vernix caseosa. Indian J Dermatol. 2008;53(2):54-60. doi: 10.4103/0019-5154.41645. PMID 19881987
- [Background] Stamatas GN, Nikolovski J, Luedtke MA, Kollias N, Wiegand BC. Infant skin microstructure assessed in vivo differs from adult skin in organization and at the cellular level. Pediatr Dermatol. 2010 Mar-Apr;27(2):125-31. doi: 10.1111/j.1525-1470.2009.00973.x. Epub 2009 Oct 4. PMID 19804498
- [Background] Suchy C, Morton C, Ramos RR, Ehrgott A, Quental MM, Burridge A, Rutledge DN. Does Changing Newborn Bath Procedure Alter Newborn Temperatures and Exclusive Breastfeeding? Neonatal Netw. 2018 Jan 1;37(1):4-10. doi: 10.1891/0730-0832.37.1.4. PMID 29436352
- [Background] Takayama JI, Teng W, Uyemoto J, Newman TB, Pantell RH. Body temperature of newborns: what is normal? Clin Pediatr (Phila). 2000 Sep;39(9):503-10. doi: 10.1177/000992280003900901. PMID 11005363
- [Background] Trevisanuto, D., & Sedin, G. （2018）. Physical environment for newborns: the thermal environment. Neonatology. A Practical Guide to Neonatal Diseases. 2nd ed. Milan: SpringerVerlag
- [Background] Verklan, M. T., & Walden, M. （2004）. Thermoregulation. In M. T. Verklan & M. Walden （Eds.）, Core curriculum for neonatal intensive care nursing （3rd ed., pp. 125-134）. St. Louis, MO: Saunders.
- [Background] Warren S, Midodzi WK, Allwood Newhook LA, Murphy P, Twells L. Effects of Delayed Newborn Bathing on Breastfeeding, Hypothermia, and Hypoglycemia. J Obstet Gynecol Neonatal Nurs. 2020 Mar;49(2):181-189. doi: 10.1016/j.jogn.2019.12.004. Epub 2020 Feb 12. PMID 32057686
- [Background] Weiner, G.M., Zaichkin, J., & Kattwinkel, J. （2016）. Textbook of neonatal resuscitation （7th ed., pp. 17-65）. Elk Grove Village, IL: American Academy of Pediatrics.
- [Background] World Health Organization. （1993）. Thermal control of the newborn: a practical guide （No. WHO/FHE/MSM/93.2）. World health organization
- [Background] World Health Organization. （1997）. Thermal protection of the newborn: a practical guide （No. WHO/RHT/MSM/97.2）. World Health Organization
- [Background] World Health Organization. （2014a）. Action plan for healthy newborn infants in the Western Pacific Region （2014-2020）. Manila: WHO Regional Office for the Western Pacific.
- [Background] WHO Recommendations on Postnatal Care of the Mother and Newborn. Geneva: World Health Organization; 2013 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK190086/ PMID 24624481
- [Background] World Health Organization. （2017）. WHO recommendations on newborn health: guidelines approved by the WHO Guidelines Review Committee （No. WHO/MCA/17.07）. World Health Organization
- [Background] World Health Organization. （2021）. Indicators for assessing infant and young child feeding practices: definitions and measurement methods. World Health Organization.
- [Result] Su Weiti (2016). To investigate the relationship between immediate postpartum skin-to-skin contact between mothers and infants, neonatal body temperature and maternal-infant emotional connection [Master's thesis, China Medical University].
- [Result] Bai DL, Wu KM, Tarrant M. Association between intrapartum interventions and breastfeeding duration. J Midwifery Womens Health. 2013 Jan-Feb;58(1):25-32. doi: 10.1111/j.1542-2011.2012.00254.x. Epub 2013 Jan 14. PMID 23317341
- [Result] Boelig RC, Manuck T, Oliver EA, Di Mascio D, Saccone G, Bellussi F, Berghella V. Labor and delivery guidance for COVID-19. Am J Obstet Gynecol MFM. 2020 May;2(2):100110. doi: 10.1016/j.ajogmf.2020.100110. Epub 2020 Mar 25. PMID 32518901
- [Result] Brown A, Jordan S. Active management of the third stage of labor may reduce breastfeeding duration due to pain and physical complications. Breastfeed Med. 2014 Dec;9(10):494-502. doi: 10.1089/bfm.2014.0048. PMID 25347567
- [Result] Chang PC, Li SF, Yang HY, Wang LC, Weng CY, Chen KF, Chen W, Fan SY. Factors associated with cessation of exclusive breastfeeding at 1 and 2 months postpartum in Taiwan. Int Breastfeed J. 2019 May 7;14:18. doi: 10.1186/s13006-019-0213-1. eCollection 2019. PMID 31080493
- [Result] Duryea EL, Nelson DB, Wyckoff MH, Grant EN, Tao W, Sadana N, Chalak LF, McIntire DD, Leveno KJ. The impact of ambient operating room temperature on neonatal and maternal hypothermia and associated morbidities: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):505.e1-505.e7. doi: 10.1016/j.ajog.2016.01.190. Epub 2016 Feb 10. PMID 26874298
- [Result] Thomi M, Pfammatter JP, Spichiger E. Parental emotional and hands-on work-Experiences of parents with a newborn undergoing congenital heart surgery: A qualitative study. J Spec Pediatr Nurs. 2019 Oct;24(4):e12269. doi: 10.1111/jspn.12269. Epub 2019 Aug 30. PMID 31468697
- [Result] Jia YS, Lin ZL, Lv H, Li YM, Green R, Lin J. Effect of delivery room temperature on the admission temperature of premature infants: a randomized controlled trial. J Perinatol. 2013 Apr;33(4):264-7. doi: 10.1038/jp.2012.100. Epub 2012 Aug 2. PMID 22858889
- [Result] Lee CC, Chiou ST, Chen LC, Chien LY. Breastfeeding-Friendly Environmental Factors and Continuing Breastfeeding Until 6 Months Postpartum: 2008-2011 National Surveys in Taiwan. Birth. 2015 Sep;42(3):242-8. doi: 10.1111/birt.12170. Epub 2015 Jun 22. PMID 26095672
- [Result] Phillips, K., DePue, L., & Mullen, S. （2020）. The effect of postpartum fatigue on exclusive breastfeeding rates at discharge: A comparison of birth methods. Journal of Comprehensive Nursing Research and Care, 5（1）, 1-5.
- [Result] Rubagumya, D., Abeid, M., Aghan, E., & Noorani, M. （2021）. Barriers to early initiation of breastfeeding in healthy neonates in an urban hospital setting. medRxiv.
- [Result] Wakamura, T., & Tokura, H. （2002）. Circadian rhythm of rectal temperature in humans under different ambient temperature cycles. Journal of thermal biology, 27（5）, 439-447.